CLINICAL TRIAL: NCT00264589
Title: Effects of an Individualized Training Program on Cardiovascular Function at Rest and During Exercise in Obese and in Type 2 Diabetic Subjects
Brief Title: Exercise Training and Cardiovascular Function in Obesity and in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHRC-I/2004/APM; DGS2005/0097 (Other: CHU Nîmes, PHRC-I competition number)
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: vascular function; cardiac function; individualized training; ultrasonography; body composition
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Population (Other): non-diabetic obese subjects and type 2 diabetic subjects
  Intervention: 8 weeks individualized training program
  Interventions: Behavioral: 8 weeks individualized training program

INTERVENTIONS:
Behavioral: 8 weeks individualized training program — no drugs added

SUMMARY:
Obesity and diabetes increase cardiovascular risk by complex and incompletely known mechanisms. The aims of this study are :

1. to compare cardiac and vascular functions at rest and during exercise in 4 groups of age-matched men, without cardiovascular diseases but exhibiting increasing cardiovascular risk: trained and untrained healthy volunteers, obese and type 2 diabetic subjects
2. to test the effects of a 8-weeks long individualized training program on these functions in obese subjects and in diabetics patients.

DETAILED DESCRIPTION:
Obesity, especially in its truncal distribution, and type 2 diabetes, increase cardiovascular risk. Mechanisms underlaying both early preclinical, and clinical cardiovascular complications are complex and still incompletely clarified.

However, relationship between central, i.e. cardiac, and peripheral, i.e. vascular dysfunctions remains unclear, as well as their respective role in reduced exercise tolerance in these populations.

Moreover, exercise training can improve both metabolic status and cardiovascular risk, and thus, has proven useful in management and prevention of chronic metabolic diseases. Nevertheless, respective effects of training on cardiac and vascular functions, and on their interaction at rest, but also during exercise, need to be clarified.

Therefore, the aims of this study are :

1. to compare cardiac and vascular functions at rest and during a local maximal leg exercise in 4 groups of age-matched men, without cardiovascular diseases but exhibiting increasing cardiovascular risk: trained and untrained healthy volunteers, obese and type 2 diabetic subjects
2. to test the effects of a 8-weeks long individualized training program on these functions in obese subjects and in diabetics patients.

ELIGIBILITY:
Inclusion Criteria:

* non-diabetic obese subjects and type 2 diabetic subjects

Exclusion Criteria:

* smoking
* known peripheral artery insufficiency
* heart failure
* uncontrolled hypertension
* thyroid disease
* insulin dependent diabetes
* for diabetics subjects : HbA1c > 10 %

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
Peripherical vascular function at rest and during exercise | before and after training
cardiac function at rest and during exercise | before and after training (8 weeks)

SECONDARY OUTCOMES:
metabolic profile (biological data) | before and after training (8 weeks)
body composition and BMI | before and after training (8 weeks)
VO2 | before and after training (8 weeks)
substrate utilization during exercise | before and after training (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Pérez-Martin, MD, PhD, Principal Investigator — University Hospital Center of Nimes
Locations (1):
- Service d'Explorations et de Médecine Vasculaire University Hospital Center, Nîmes, Nimes, France

REFERENCES:
- [Result] Vinet A, Karpoff L, Walther G, Startun A, Obert P, Goret L, Dauzat M, Perez-Martin A. Vascular reactivity at rest and during exercise in middle-aged obese men: effects of short-term, low-intensity, exercise training. Int J Obes (Lond). 2011 Jun;35(6):820-8. doi: 10.1038/ijo.2010.206. Epub 2010 Sep 28. PMID 20877288